CLINICAL TRIAL: NCT00098436
Title: A Phase I Study Of Cloretazine™ (VNP40101M) And Temozolomide In Patients With Hematologic Malignancies
Brief Title: Temozolomide and VNP40101M in Treating Patients With Relapsed or Refractory Leukemias
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: VION-CLI-036; CDR0000405825 (Registry Identifier: PDQ (Physician Data Query)); CWRU-050419
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2008-08

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; blastic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis; Congenital Abnormalities | interventions — laromustine; Temozolomide

INTERVENTIONS:
Drug: laromustine
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide and VNP40101M, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Temozolomide may also help VNP40101M kill more cancer cells by making cancer cells more sensitive to the drug. Giving temozolomide together with VNP40101M may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of temozolomide and VNP40101M in treating patients with relapsed or refractory leukemias.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of temozolomide and VNP40101M in patients with relapsed or refractory leukemias.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Patients receive oral temozolomide twice daily on days 1-3 (for 5 doses) followed by VNP401010M IV over 15-60 minutes on day 3 (course 1). Patients achieving a complete or partial response or having ≥ 50% reduction in bone marrow blasts may receive a second course of therapy no earlier than day 43. Courses may be repeated approximately every 6 weeks at the discretion of the sponsor and in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of temozolomide until a dose that depletes leukemic blast AGT in at least 4 of 6 patients is determined. Once this dose is determined, cohorts of 3-6 patients receive escalating doses of VNP401010M until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 10 patients are treated at the MTD.

PROJECTED ACCRUAL: Approximately 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Acute myeloid leukemia
  * Acute lymphoblastic leukemia
  * Chronic myelogenous leukemia in blast crisis
* Relapsed or refractory disease
* No known standard therapy that is anticipated to result in a durable remission exists
* CNS leukemia allowed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT or AST ≤ 3 times ULN
* Chronic hepatitis allowed

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* No active heart disease, including any of the following:

  * Myocardial infarction within the past 3 months
  * Symptomatic coronary artery disease
  * Arrhythmias not controlled by medication
  * Uncontrolled congestive heart failure

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No uncontrolled active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Concurrent hydroxyurea allowed within the first 10 days of study drug administration for control of elevated blast levels or platelet counts

  * Maximum hydroxyurea dose 5 g daily
* No persistent chronic toxic effects from prior chemotherapy > grade 1

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Recovered from all prior therapy
* At least 2 weeks since prior myelosuppressive cytotoxic agents (in the absence of rapidly progressive disease)
* No more than 2 leukapheresis procedures within the first 10 days of study drug administration for control of elevated blast levels or platelet counts
* No concurrent disulfiram
* No other concurrent anticancer drugs
* No other concurrent standard or investigational treatment for leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2004-09; Primary Completion 2006-10 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonny L. Johnson, RN, MSN, Study Chair — Vion Pharmaceuticals
Locations (4):
- United States (4):
  - American Health Network - North Illinois Street, Indianapolis, Indiana
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio

REFERENCES:
- [Result] Rizzieri D, LoRusso S, Tse W, Khan K, Advani A, Moore J, Karsten V, Cahill A, Gerson SL. Phase I study of temozolomide and laromustine (VNP40101M) in patients with relapsed or refractory leukemia. Clin Lymphoma Myeloma Leuk. 2010 Jun;10(3):211-6. doi: 10.3816/CLML.2010.n.033. PMID 20511167